CLINICAL TRIAL: NCT05002153
Title: The Role of Microbiome in Recurrent Obesity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assaf Harofeh MC (Other Government)
Collaborators: Weizmann Institute of Science (Other)
Responsible Party: Sponsor-Investigator, Assaf Harofeh MC, Principal Investigator, Assaf-Harofeh Medical Center
Organization: Assaf-Harofeh Medical Center (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0215-19-ASF; NCT04697550 (obsolete NCT alias)
Record Dates: First submitted 2021-07-27; First posted 2021-08-12 (Actual); Last update posted 2021-12-28 (Actual); Status verified 2021-12

CONDITIONS: Obesity; Weight Loss; FMT
MeSH Terms: conditions — Obesity; Weight Loss | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fecal Microbiota Transplantation (FMT) (Experimental): FMT capsules administration - intervention arm
  Interventions: Other: Fecal microbiota transplantation (FMT)
- Placebo (Placebo Comparator): Placebo capsules administration
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Fecal microbiota transplantation (FMT) — FMT is the process of transferring stool from a healthy donor to another.
  Arms: Fecal Microbiota Transplantation (FMT)
Other: Placebo — Placebo capsules consist a combination of agarose in normal saline/glycerol (the same vehicle as in a FMT capsules)
  Arms: Placebo

SUMMARY:
This past century witnessed a significant increase in the prevalence of obesity, when since 1980 worldwide obesity has more than doubled. According to the World Health Organization, 39% of adults from the age of 18 years or older are overweight while 13% are obese. Successful maintenance of weight loss as losing at least 10% of the initial body weight and maintaining it for at least one year. However, keeping the low body weight is rarely maintained, as 80% of people who lost 10% of their body weight will return to their initial weight within a year. When weight loss is maintained for 2-5 years the chance of long term success was shown to dramatically increase.

Although there is no agreement as to what contributes to the recurrent weight regain phenomenon (also known as 'weight cycling' or 'yo-yo diet'), it is strongly associated with the risk of developing metabolic risk factors and their complications including heart disease and all-cause mortality.

Altering the gut microbiota is one method to treat disease states associated with gut bacteria. For instance, fecal microbiota transplant (FMT) or fecal bacteriotherapy, is the process of transferring stool from a healthy donor to another. The goal of FMT is to restore host health by increasing diversity and function of the gut microbiota. The main advantage of FMT over probiotics is its ability to transplant the entire gut microbiota and metabolites from the donor to the recipient.

Although numerous individual microbes have been identified as related to obesity, multiple studies suggest that loss of microbial diversity has a stronger impact on the development of metabolic dysfunction, this diversity may be restored by FMT.

This study will determine whether microbiome modulation might be a possible future target against recurrent obesity in humans, and whether orally administered FMT from a lean donor, post weight loss might be an effective intervention to prevent weight regain.

DETAILED DESCRIPTION:
This is a placebo-controlled, double blinded interventional study evaluating high intensity oral fecal microbiota transplantation from lean healthy donors to prevent weight regain after a successful weight loss intervention. Volunteers will be recruited in the following ways: e-mail, and social media. Volunteers wishing to participate will be asked to complete a questionnaire regarding the aforementioned inclusion and exclusion criteria. Volunteers who qualify for the study will be invited to an introductory meeting at the Weizmann Institute of Science. The details of the experiment and potential risks or discomforts involved in it will be presented, after which the volunteers will sign informed consent forms. Volunteers will start the study and become active participants for a maximal duration of two years, depending on the weight loss process.

The study will comprise of four parts:

1. Baseline - one week of profiling and screening.
2. Nutritional intervention - weight loss intervention which will be based on Mediterranean hypocaloric diet restriction. Meetings will occur twice a month starting from the second week of the study for a three-month period.
3. FMT/ Placebo intervention - 5 weekly cycles of high intensity lean donor FMT/placebo will be administered starting after reaching a weight loss of 5 to 10% of total body weight. Each cycle will consist of 10 capsules administered on two consecutive days (total 100 capsules)
4. Follow-up meetings - total follow up of one year after FMT cycles. Meetings will occur every month for the first 3 months of the study, and every 3 months, Afterwards.

ELIGIBILITY:
Inclusion Criteria:

* 28<BMI>35
* Age: 18-65
* Capable of working with a smartphone application

Exclusion Criteria:

* Consumption of antibiotics/probiotics/oral antifungals 3 months prior to the first day of the experiment.
* Pregnancy, fertility treatments, breastfeeding women six months prior to enrollment and during the study.
* Chronic disease (e.g. AIDS, Cushing syndrome, CKD, acromegaly, hyperthyroidism/hypothyroidism etc.)
* Cancer and recent anticancer treatment
* Psychiatric disorders
* Coagulation disorders
* IBD (inflammatory bowel diseases)
* Bariatric surgery
* Eating disorders (Anorexia nervosa. Bulimia nervosa. Binge eating disorder, Night eating syndrome).
* Alcohol or substance abuse
* Weight loss attempts one year prior to the first day of the experiment - independent or with a dietitian.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-01 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Microbiome Profiling | 1.5 years
  Collection of stool, urine and oral samples for microbiome composition. 16S RNA analysis.
Reaching Target Weight | 1.5 years
  Investigate the effect of FMT administration after reaching target weight (kg) on the recurrent weight regain phenomenon.

SECONDARY OUTCOMES:
Glycemic Response | 1.5 years
  Performing continuous glucose monitoring (CGM) and oral glucose tolerance test (OGTT)
Metabolic Rate | 1.5 years
  RMR
Substrate Utilization | 1.5 years
  measured by indirect calorimetry

CONTACTS AND LOCATIONS:
Overall Officials: Ilan Youngster, Dr., Principal Investigator — Asaf Harofe Medical Center, Be'er Yaacov, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wing RR, Phelan S. Long-term weight loss maintenance. Am J Clin Nutr. 2005 Jul;82(1 Suppl):222S-225S. doi: 10.1093/ajcn/82.1.222S. PMID 16002825
- [Background] Mackie GM, Samocha-Bonet D, Tam CS. Does weight cycling promote obesity and metabolic risk factors? Obes Res Clin Pract. 2017 Mar-Apr;11(2):131-139. doi: 10.1016/j.orcp.2016.10.284. Epub 2016 Oct 20. PMID 27773644
- [Background] Wing RR, Hill JO. Successful weight loss maintenance. Annu Rev Nutr. 2001;21:323-41. doi: 10.1146/annurev.nutr.21.1.323. PMID 11375440
- [Background] Bangalore S, Fayyad R, Laskey R, DeMicco DA, Messerli FH, Waters DD. Body-Weight Fluctuations and Outcomes in Coronary Disease. N Engl J Med. 2017 Apr 6;376(14):1332-1340. doi: 10.1056/NEJMoa1606148. PMID 28379800
- [Background] Lee P, Yacyshyn BR, Yacyshyn MB. Gut microbiota and obesity: An opportunity to alter obesity through faecal microbiota transplant (FMT). Diabetes Obes Metab. 2019 Mar;21(3):479-490. doi: 10.1111/dom.13561. Epub 2018 Nov 20. PMID 30328245
- [Background] Thaiss CA, Itav S, Rothschild D, Meijer MT, Levy M, Moresi C, Dohnalova L, Braverman S, Rozin S, Malitsky S, Dori-Bachash M, Kuperman Y, Biton I, Gertler A, Harmelin A, Shapiro H, Halpern Z, Aharoni A, Segal E, Elinav E. Persistent microbiome alterations modulate the rate of post-dieting weight regain. Nature. 2016 Dec 22;540(7634):544-551. doi: 10.1038/nature20796. Epub 2016 Nov 24. PMID 27906159
- See also: World Health Organization. WHO Obesity and Overweight — http://www.who.int/mediacentre/factsheets/fs311/en/.